CLINICAL TRIAL: NCT03486587
Title: A Single-arm, Single-institutional, Phase II Study Evaluating the Efficacy and Safety of Bacillus Cereus (Changfukang®) in the Prevention of Afatinib-associated Diarrhea in NSCLC Patients
Brief Title: A Study Evaluating Bacillus Cereus in the Prevention of Afatinib-associated Diarrhea
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Participants have better treatment selection, resulting in a slow recruitment.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-FXY-137
Record Dates: First submitted 2018-03-18; First posted 2018-04-03 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Diarrhea; Treatment Side Effects
Keywords: afatinib; diarrhea; Bacillus Cereus; NSCLC
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Intervention Model Description: a single-arm, single-institutional, phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Changfukang® group (Experimental): Patients in Changfukang group will receive Changfukang® (Bacillus Cereus tablets).
  Interventions: Drug: Bacillus Cereus tablets

INTERVENTIONS:
Drug: Bacillus Cereus tablets — Bacillus Cereus tablets was taken two tablets three times a day.

SUMMARY:
Afatinib is an irreversible ErbB-family blocker with approved clinical activity in non-small-cell lung cancer (NSCLC) with EGFR mutations. It has received regulatory approval for use as a treatment for patients with lung adenocarcinoma whose tumors harbour activating EGFR mutations within exons 18-21 of the EGFR receptor, or patients with lung squamous cell carcinoma whose disease progress after platinum-based doublet chemotherapy. However, diarrhea is the most commonly reported adverse events associated with afatinib treatment (> 90%). Although these events are generally mild to moderate in severity, diarrhea adversely affects the tolerability of cancer treatment, and in severe cases diarrhea has the potential to affect the efficacy of treatment due to poor compliance, or treatment interruption, or dosage reduction. Currently, no prophylactic measure was demonstrated efficaciously. Bacillus cereus is an aerobic spore-forming bacterium that is commonly found in soil. The efficacy of Bacillus cereus in the management of afatinib treatment-associated diarrhoea has not been extensively evaluated in clinical studies. This is a single-arm, single-institutional, phase II study evaluating the efficacy and safety of Bacillus cereus (Changfukang®) in the prevention of afatinib-associated diarrhea in NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastastic non-small-cell lung cancer
* Suitable for the treatment of afatinib assessed by investigator
* Age >=18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy of at least 12 weeks
* Able to swallow and retain oral medications
* Women of childbearing potential must agree and commit to the use of a highly effective non-hormonal method of contraception, ie, intrauterine device, bilateral tubal ligation, vasectomized partner, or abstinence (only when it is the preferred lifestyle of the patient), from the time of informed consent until 28 days after the last dose of the investigational products. Men and their female partners of childbearing potential must agree and commit to use a highly effective method of contraception (ie, any of the above methods or hormonal contraception associated with inhibition of ovulation) while on treatment and for 3 months after last dose of investigational products
* Provide written, informed consent to participate in the study and follow the study procedures
* Patient has adequate bone marrow as defined by the following laboratory values:

  * White blood cell ≥ 3.0 × 109/L
  * Absolute neutrophil count ≥ 1.5 × 109/L
  * Platelets ≥ 75 × 109/L
* Patient has adequate organ function as defined by the following laboratory values:

  * In absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) should be below 2.5 × ULN. If the patient has liver metastases, ALT and AST should be < 5 × ULN
  * Total serum bilirubin < ULN; or total bilirubin ≤ 3.0 × ULN with direct bilirubin within normal range of the central laboratory in patients with well documented
  * Gilbert's Syndrome
  * Serum creatinine ≤ 1.5 × ULN

Exclusion Criteria:

* Previous treatment with EGFR-TKI or anti-EGFR antibody
* History of gastrointestinal disease with diarrhea as the primary symptom in the last three months.
* Another malignancy within 3 years prior to randomization, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, basal or squamous cell carcinoma or non-melanomatous skin cancer
* Diagnosed as having CNS metastases, except those whose CNS disease were stable and dehydration treatment were unrequired within 4 weeks prior to the first dose of afatinib
* Any severe and / or uncontrolled medical conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Diarrhoea rate of all grades | Up to 4 weeks
  Proportion of subjects experiencing diarrhoea of all grades, as defined by the National Cancer Institute common terminology criteria for adverse events (NCI CTCAE) version 4.03, recorded as AEs in the Electronic case report form (eCRF)

SECONDARY OUTCOMES:
Diarrhoea rate of grade 2 and above | Up to 4 weeks
  Proportion of subjects experiencing diarrhoea of grade 2 and above, as defined by the NCI CTCAE, version 4.03 and recorded as AEs in the eCRF
Diarrhoea rate of grade 3 and above | Up to 4 weeks
  Proportion of subjects experiencing diarrhoea of grade 3 and above, as defined by the NCI CTCAE, version 4.03 and recorded as AEs in the eCRF
Days of diarrhoea of all grades | Up to 4 weeks
  Number of days of subjects experiencing diarrhoea of all grades, as defined by the NCI CTCAE, version 4.03 and recorded as AEs in the eCRF
Days of diarrhoea of grade 2 and above | Up to 4 weeks
  Number of days of subjects experiencing diarrhoea of grade 2 and above, as defined by the NCI CTCAE, version 4.03 and recorded as AEs in the eCRF
Days of diarrhoea of grade 3 and above | Up to 4 weeks
  Number of days of subjects experiencing diarrhoea of grade 3 and above, as defined by the NCI CTCAE, version 4.03 and recorded as AEs in the eCRF
Proportion of subjects taking anti-diarrheal medication | Up to 4 weeks
  Proportion of subjects taking anti-diarrhoeal medication as recorded in the eCRF
Proportion of subjects with AEs and SAEs | Up to 4 weeks
  Proportion of subjects with AEs and SAEs were assessed from the start of the study until end of study as recorded in the eCRF

OTHER OUTCOMES:
Overall Response Rate | Up to 4 weeks
  Overall response rate as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1
Clinical Benefit Response | Up to 4 weeks
  Clinical benefit response as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1
Progression-free Survival | Up to 4 weeks
  Progression-free Survival as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided